CLINICAL TRIAL: NCT04850833
Title: Post-operative Functional Disability in Unrecognized Cognitive Impairment (POF) Study: an Observational Cohort Study in Patients Undergoing Non-cardiac Surgery
Brief Title: Post-operative Functional Disability in Unrecognized Cognitive Impairment (POF) Study
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 20-6186
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Impairment (CI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective multicenter cohort study, which will determine the prevalence of preoperative cognitive impairment (CI) using the Modified Telephone Interview for Cognitive Status (TICS-M), Eight-items interview to Differentiate Aging and Dementia (AD8), Telephone Montreal Cognitive Assessment (T-MoCA), and a single cognitive question from the Centers for Disease Control and Prevention (CDC). We would also determine the (1) the degree of agreement in screening results between each cognitive screening tool, (2) risk factors associated with screening positive for CI on each tool, and (3) the prevalence and/or trajectory of postoperative delirium, sleep disturbances, functional disability, instrumental activities of daily living (IADL), depression, quality of health, frailty, and pain in older surgical patients and its association with CI. This study will target older patients from the pre-operative clinics at Toronto Western Hospital and Mount Sinai Hospital (MSH), Toronto. Research staff will identify eligible patients who are scheduled for elective non-cardiac surgery. Written informed consent to participate in the study will be obtained from all patients.

DETAILED DESCRIPTION:
The primary aim of this study is to (1) determine the prevalence of CI preoperatively in older surgical adults using virtual or telephone cognitive instruments, (2) determine the degree of agreement in screening results between each cognitive screening tool, and (3) explore the prevalence and trajectory of preoperative and postoperative outcomes and its association with CI. The outcomes include functional disability, IADL, sleep disturbances, quality of health, frailty, pain and depression.

In a preoperative assessment 1-30 days prior to their scheduled surgery, patients will be asked via telephone to complete TICS-M and T-MoCA and an online questionnaire, including the AD8, CDC single cognitive question, World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0), IADL, EuroQol 5 Dimension (EQ-5D-5L), Geriatric Depression Scale (GDS), 5-item FRAIL questionnaire, (FRAIL), visual analog pain scale (VAS pain), Single-item Sleep Quality Scale (SQS), Pittsburgh Sleep Quality Index (PSQI), and STOP questionnaire. These questionnaires will be repeated at follow-up visits at 30-, 90-, and 180-days post-surgery. At the hospital on post-operatively days 1-3, the Confusion Assessment Method (CAM), SQS, and VAS pain will be administered during the in-person visit. Chart review of delirium will also be conducted during patients' stay at the hospital.

ELIGIBILITY:
Major Inclusion Criteria:

* patients ≥ 65 years old;
* patients scheduled for elective non-cardiac surgery
* able to be contacted by telephone for follow up.

Major Exclusion Criteria:

* patients with previous dementia diagnosis,
* patients scheduled for outpatient surgery,

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients scheduled to undergo elective inpatient non-cardiac surgery under general and/ or regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of cognitive impairment via remote (virtual/telephone) assessment | Pre-surgery, 30-, 90- and 180-days post-surgery
  Prevalence of cognitive impairment via remote (virtual/telephone) assessment as detected by the TICS-m (modified telephone interview for cognitive status). The TICS-m is scored from 0-50 with a score of 31 or below indicating cognitive impairment.
Prevalence of cognitive impairment via remote (virtual/telephone) assessment | Pre-surgery, 30-, 90- and 180-days post-surgery
  Prevalence of cognitive impairment via remote (virtual/telephone) assessment as detected by the T-MoCA (telephone Montreal cognitive assessment). The T-MoCA is scored from 0-22 with a score of 18 or below indicating cognitive impairment.
Prevalence of cognitive impairment via remote (virtual/telephone) assessment | Pre-surgery, 30-, 90- and 180-days post-surgery
  Prevalence of cognitive impairment via remote (virtual/telephone) assessment as detected by the AD8 (eight-item interview to differentiate aging and dementia). The AD8 is scored from 0-8 with a score of two or more indicating cognitive impairment.
Prevalence of cognitive impairment via remote (virtual/telephone) assessment | Pre-surgery, 30-, 90- and 180-days post-surgery
  Prevalence of cognitive impairment via remote (virtual/telephone) assessment as detected by the CDC Single Cognitive Question. The CDC Single Cognitive Question is a yes/no question where answers of yes indicate cognitive impairment.
Degree of agreement in screening results (Cohen's Kappa (κ) coefficients) | Pre-surgery
  The degree of agreement in screening results among the screening tools by calculating Cohen's Kappa (κ) coefficients.
The trajectories and prevalence or incidence of patient-reported outcomes | Pre-surgery, 30-, 90- and 180-days post-surgery
  The trajectories and prevalence or incidence of functional disability as measured through the WHODAS 2.0 (World Health Organization Disability Assessment Schedule 2.0) in participants with vs without preoperative functional disability and in participants with vs without CI. A five-point rating scale is used for each question (none = 0, mild = 1, moderate = 2, severe = 3, extreme/cannot do = 4), and a higher WHODAS score indicates greater disability.
The trajectories and prevalence or incidence of patient-reported outcomes | Pre-surgery, 30-, 90- and 180-days post-surgery
  The trajectories and prevalence or incidence of instrumental activities of daily living (IADL) as measured through the IADL in participants with CI vs those without. It is scored from 0-8 where a higher score indicates high function and independence.
The trajectories and prevalence or incidence of patient-reported outcomes | Pre-surgery, 30-, 90- and 180-days post-surgery
  The trajectories and prevalence or incidence of sleep disturbances as measured through the PSQI (Pittsburgh Sleep Quality Index) in participants with CI vs those without. It is scored from 0-21 where a higher score indicates worse sleep quality.
The trajectories and prevalence or incidence of patient-reported outcomes | Pre-surgery, 30-, 90- and 180-days post-surgery
  The trajectories and prevalence or incidence of sleep quality as measured through the SQS (Single-Item Sleep Quality Scale) in participants with CI vs those without. It is scored from 0-10 where a higher score indicates better sleep quality.
The trajectories and prevalence or incidence of patient-reported outcomes | Pre-surgery, 30-, 90- and 180-days post-surgery
  The trajectories and prevalence or incidence of depression as measured through the GDS (Geriatric Depression Scale) in participants with vs without preoperative depression and in participants with vs without CI. It is scored from 0-15 where a higher score indicates depression.
The trajectories and prevalence or incidence of patient-reported outcomes | Pre-surgery, 30-, 90- and 180-days post-surgery
  The trajectories and prevalence or incidence of pain as measured through the VAS Pain (Visual Analog Scale for Pain) in participants with CI vs those without. It is scored from 0-10 where a lower score indicates worse pain.
The trajectories and prevalence or incidence of patient-reported outcomes | Pre-surgery, 30-, 90- and 180-days post-surgery
  The trajectories and prevalence or incidence of frailty as measured through the 5-item FRAIL questionnaire (Fatigue, resistance, ambulation, illnesses, and loss of weight) in participants with vs without preoperative frailty and in participants with vs without CI. It is scored from 0-5 where higher scores indicate frailty.
The trajectories and prevalence or incidence of patient-reported outcomes | Pre-surgery, 30-, 90- and 180-days post-surgery
  The trajectories and prevalence or incidence of quality of health as measured through the EQ5D5L (EuroQol 5 Dimension) in participants with CI vs those without. Each dimension on the tool has five response levels and one level from each dimension is combined to give a health state ranging from 11111 (full health) to 55555 (worst health). The health states are converted into a single index utility where lower values indicate worse quality of health

SECONDARY OUTCOMES:
The incidence of postoperative delirium post-surgery | Post-op day 1-3
  The incidence of postoperative delirium as measured by the Confusion Assessment Method (CAM) conducted by the research and nursing team and medical chart review.
Discharge destination of participants from chart review post-surgery | Post-op day 1-3
  Discharge destination (assess where the participant will be discharged to once out of hospital up to 30-days post-op)
Hospital length of stay (LOS) of participants post-surgery | Post-op day 1-3
  Hospital length of stay
Days spent at home (DAH30) of participants post-surgery | 30-days post-surgery
  DAH30 (days spent at home) at 30 days post-surgery
Mortality (number of participants who have died) post-surgery | 30-, 90- and 180-days post-surgery
  Mortality
Number of participants who have been re-admitted to the hospital post-surgery | 30-, 90- and 180-days post-surgery
  Hospital re-admission
Number of participants who have visited the emergency department post-surgery | 30-, 90- and 180-days post-surgery
  Emergency department visit
Incidence of postoperative complications of participants post-surgery | 30-, 90- and 180-days post-surgery
  All-cause postoperative complications
Incidence of re-operation or revision surgery post-surgery | 30-, 90- and 180-days post-surgery
  Re-operation or revision surgery
Risk factors for screening positive on each cognitive screening tool | Pre-surgery
  Preoperative risk factors associated with screening positive on each cognitive screening tool

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS MD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - 399 Bathurst St., Toronto Western Hospital, Dept. of Anesthesia, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Lu YT, Yan E, Alhamdah Y, Kapoor P, Lovblom LE, Saripella A, Wong J, Chung F. The prevalence and trajectory of frailty in older surgical patients: A longitudinal multicentre cohort study. Anaesth Crit Care Pain Med. 2025 Sep;44(5):101582. doi: 10.1016/j.accpm.2025.101582. Epub 2025 Jun 27. PMID 40582463